CLINICAL TRIAL: NCT06669078
Title: A Prospective, Open, Randomized Controlled, Multicenter, Exploratory Clinical Study of NALIRIFOX Combined With PD-1 Sequential Radiotherapy Versus NALIRIFOX for Conversion Therapy for Locally Advanced Pancreatic Cancer
Brief Title: NALIRIFOX Combined With PD-1 Sequential Radiotherapy Versus NALIRIFOX as Conversion Therapy of Locally Advanced Pancreatic Cancer
Acronym: NALIRIFOX
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-PC-JS06
Record Dates: First submitted 2024-10-27; First posted 2024-11-01 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced Pancreatic Cancer
Keywords: NALIRIFOX; Conversion Therapy; Locally Advanced Pancreatic Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NALIRINOX combined with PD-1 synchronous sequential SBRT group (Experimental): Nal-IRI+Oxaliplatin+5- FU +PD-1, these drugs are given on d1, d15, 28 days as one cycle, SBRT is performed during the third and fourth cycle.
  Interventions: Drug: Nal-lRl+Oxaliplain+5- FU +PD 1
- NALIRIFOX group (Experimental): Nal-IRI+Oxaliplatin+5- FU, these drugs are given on d1, d15, 28 days as one cycle.
  Interventions: Drug: Nal-lRl+Oxaliplain+5- FU

INTERVENTIONS:
Drug: Nal-lRl+Oxaliplain+5- FU +PD 1 — Nal-lRl+Oxaliplatin+5- FU +PD-1, these drugs are given on d1, d15, 28 days as one cycle, SBRT is performed during the third and fourth cycle.
  Arms: NALIRINOX combined with PD-1 synchronous sequential SBRT group
Drug: Nal-lRl+Oxaliplain+5- FU — Nal-lRl+Oxaliplatin+5- FU, these drugs are given on d1, d15, 28 days as one cycle.
  Arms: NALIRIFOX group

SUMMARY:
The purpose of the prospective, open, randomized controlled, multicenter, exploratory clinical study is to evaluate efficacy and safety of NALIRIFOX Combined With PD-1 Sequential Radiotherapy Versus NALIRIFOX for Conversion Therapy for Locally Advanced Pancreatic Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confi rmed pancreatic cancer;
2. ECOG performance no more than 1;
3. Radiographically assessed as locally advanced pancreatic cancer according ;
4. No previous anti-tumor therapy;
5. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. Prior anti-tumor therapy of any kind;
2. Known to be symptomatic central nervous system metastasis and/or cancerous meningitis.
3. Patients with autoimmune disease or immune deficiency who are treated with immuno-suppressive drugs;
4. Patients with bleeding tendency;
5. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-10-30 (Estimated); Primary Completion 2027-10-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
1 year OS rate | Up to 12 months]
  Proportion of patients alive from randomization to 1 year

SECONDARY OUTCOMES:
R0/R1 rate | Up to 6 months
  Percentage of patients who achieved R0/RI resection
The rate of mPR | Up to 6 months
  Proportion of patients who achieved mPR by post-operative specimen testing
OS | Up to 24 months
  Time from randomization to death
ORR | Up to 6 months
  According to RECIST version 1.1, the proportion of patients who achieved remission (PR+CR) after treatment and maintained the minimum time-frame requirement.
PFS | Up to 12 months
  Time from randomization to disease progression and/or death.
Surgical resection rate | Up to 6 months
  Operable rate
The incidence of grade 3 or higher AE and serious adverse event(SAE) [Safety] | From the first treatment to 28 days after the last treatment, about 6 months
  Using the Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0, we analyzed the data of all subjects who received at least one study treatment. We collected and summarized the overall incidence of adverse events (AE), the incidence of grade 3 or higher AE, and the incidence of serious adverse events (SAE).

IPD SHARING:
Plan to Share IPD: No